CLINICAL TRIAL: NCT00943891
Title: A Study of Lymphangiogenesis in Colorectal and Nasopharyngeal Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National University Hospital, Singapore (Other)
Other Study IDs: MC01/09/08
Record Dates: First submitted 2009-07-20; First posted 2009-07-22 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Colorectal Cancer; Nasopharyngeal Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Nasopharyngeal Neoplasms

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — CRC and NPC tumor specimens will be obtained.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Tumor biopsies
  Interventions: Procedure: Tumor biopsies

INTERVENTIONS:
Procedure: Tumor biopsies

SUMMARY:
1. To determine the association between LVD and clinico-pathologic variables in archived colorectal cancer and Nasopharyngeal carcinoma specimens
2. To determine the association between VEGF-C,-D expression with COX-2 expression and clinico-pathologic variables in colorectal cancer and Nasopharyngeal carcinoma
3. To determine the effect of celecoxib on lymphangiogenesis in Nasopharyngeal carcinoma Lymphangiogenesis and factors modulating lymphangiogenesis are associated with clinico-pathological outcome in Nasopharyngeal carcinoma and colorectal cancer. Celecoxib down-regulates lymphangiogenesis Archival colorectal cancer and Nasopharyngeal carcinoma tumor specimens will be obtained from the Department of Pathology. To determine the effect of celecoxib on lymphangiogenesis in Nasopharyngeal carcinoma, the investigators intend to analyze archived specimens collected in a previously conducted study. Colorectal tumor and nodal specimens and Nasopharyngeal carcinoma primary will be examined for MVD, LVD and growth factor expression using established haematoxylin and eosin and immunohistochemical techniques. Quantification of LVD and MVD shall be performed by two pathologists blinded to clinico-pathological variables using standardised methods.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients are eligible
* Patients 21 years or older

Exclusion Criteria:

* None

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Colorectal and nasopharyngeal cancer.
Sampling Method: Non-Probability Sample
Enrollment: 500
Dates: Start 2008-07; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ross Andrew Soo, MBBS, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Background] Stacker SA, Caesar C, Baldwin ME, Thornton GE, Williams RA, Prevo R, Jackson DG, Nishikawa S, Kubo H, Achen MG. VEGF-D promotes the metastatic spread of tumor cells via the lymphatics. Nat Med. 2001 Feb;7(2):186-91. doi: 10.1038/84635. PMID 11175849
- [Background] Mandriota SJ, Jussila L, Jeltsch M, Compagni A, Baetens D, Prevo R, Banerji S, Huarte J, Montesano R, Jackson DG, Orci L, Alitalo K, Christofori G, Pepper MS. Vascular endothelial growth factor-C-mediated lymphangiogenesis promotes tumour metastasis. EMBO J. 2001 Feb 15;20(4):672-82. doi: 10.1093/emboj/20.4.672. PMID 11179212